CLINICAL TRIAL: NCT01340950
Title: Clinical Trial of CNS Penetrating ART to Prevent NeuroAIDS in China
Brief Title: Clinical Trial of Brain-Penetrating HIV Drugs to Prevent Cognitive Impairment in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); National Center for AIDS/STD Control and Prevention, China CDC (Other Government); Beijing YouAn Hospital (Other); Beijing Ditan Hospital (Other); Peking University (Other)
Responsible Party: Principal Investigator, Scott Letendre, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH092225 (NIH); 1R01MH092225-01 (NIH)
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infections; Central Nervous System Diseases; Dementia
Keywords: Prevention; Anti-Retroviral Agents; Neuropsychological Tests
MeSH Terms: conditions — HIV Infections; Central Nervous System Diseases; Dementia | interventions — Zidovudine; Lamivudine; Nevirapine; efavirenz, lamivudine, tenofovir disoproxil fumarate drug combination; Tenofovir; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Better-Penetrating ART (Active Comparator): zidovudine 300 mg orally every 12 hours lamivudine 300 mg orally daily nevirapine 200 mg orally every 12 hours
  Interventions: Drug: zidovudine-lamivudine-nevirapine
- Worse-Penetrating ART (Active Comparator): tenofovir disoproxil fumarate 300 mg orally daily lamivudine 150 mg orally every 12 hours efavirenz 600 mg orally daily
  Interventions: Drug: tenofovir-lamivudine-efavirenz

INTERVENTIONS:
Drug: zidovudine-lamivudine-nevirapine — 96 weeks of zidovudine 300 mg orally twice daily, lamivudine 300 mg orally daily, nevirapine 200 mg orally daily for the first 14 days then 200 mg orally twice daily
  Other Names: Retrovir, Epivir, Viramune
  Arms: Better-Penetrating ART
Drug: tenofovir-lamivudine-efavirenz — 96 weeks of tenofovir disoproxil fumarate 300 mg orally daily, lamivudine 300 mg orally daily, efavirenz 600 mg orally daily
  Other Names: Viread, Epivir, Sustiva
  Arms: Worse-Penetrating ART

SUMMARY:
This primary aim of the project is to determine the association between antiretroviral therapy that better distributes into the central nervous system and prevention of HIV-associated neurocognitive impairment.

DETAILED DESCRIPTION:
Advances in treatment have transformed HIV disease to a chronic illness in most individuals in the U.S. The most common central nervous system (CNS) complication of chronic HIV disease is HIV-associated neurocognitive disorder (HAND). In the U.S., HAND prevalence estimates range up to 55% of treated individuals. HAND is also common outside the U.S. For example, our prior project in China identified that more than a third of nearly 150 treated HIV(+) individuals in Anhui and Yunnan provinces had HAND. Data such as these support that the benefits of antiretroviral therapy (ART) can be incomplete, with many patients not returning to normal neurocognitive performance or, worse, developing new neurocognitive impairment while taking ART.

One explanation for this is the limited penetration of some antiretrovirals into the nervous system. Recent reports have identified that worse antiretroviral penetration characteristics are associated with worse control of HIV replication and worse neurocognitive performance. Most reports, however, have focused on treatment - rather than prevention - of HAND. Like many other medical conditions, prevention of HAND may be a more cost-effective public health goal than treating disease that has already occurred.

We are building on our prior work in China by performing a phase 4, randomized, controlled clinical trial of the safety and effectiveness of ART that differs in its penetration characteristics in 250 ART-naive individuals who have normal neurocognitive performance. The primary objective will be to determine the effects of better penetrating (BP) ART (zidovudine-lamivudine-nevirapine) compared with worse penetrating (WP) ART (tenofovir-lamivudine-efavirenz) on the prevention of HAND. We hypothesize that volunteers who are randomized to BP-ART will be less likely to neurocognitively decline over 96 weeks of observation than those who are randomized to WP-ART. The secondary objective will be to assess the influence on study outcomes of two conditions: persistent immune activation and viral hepatitis. In an exploratory aim, the project will also assess the influence on study outcomes of a concise panel of drug disposition-associated genetic polymorphisms.

Demonstrating that HAND can be prevented by using BP-ART should influence HIV treatment guidelines in the U.S., China, and elsewhere and ultimately lead to preservation of normal neurocognitive functioning in people afflicted with HIV/AIDS.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of at least 18 years of age.
* Ability and willingness of subject to give written informed consent.
* HIV-1 infection, as documented by enzyme-linked immunosorbent assay (ELISA) and confirmed by Western blot at any time prior to study entry. Plasma HIV-1 RNA is acceptable as an alternative confirmatory test.
* Antiretroviral drug-naïve, defined as ≤10 days of ART at any time prior to entry.
* Clinical HIV-1 RNA ≥1000 copies/mL obtained within 90 days of study screening.
* Clinical blood CD4+ cell count < 350/mm3 (for men) or <250/mm3 (for women) within 60 days of study screening.
* Performance within the expected normal range on the project's comprehensive, standardized battery of neuropsychological tests within 4 weeks.
* For women of child-bearing potential (WOCBP), negative serum or urine pregnancy test at screening and within 48 hours prior to initiating study medications.

Exclusion Criteria:

* Serious illness requiring systemic treatment or hospitalization within 4 weeks.
* Unacceptable laboratory values obtained within 4 weeks prior to study entry.
* Untreated syphilis.
* Child Pugh Class C hepatic impairment.
* Active Hepatitis B Virus infection.
* Known allergy/sensitivity to study drugs or their formulations.
* Severe or untreated conditions that could affect NP test performance.
* Such conditions include but are not limited to current substance use disorder, poorly controlled diabetes, uncontrolled seizure disorder, and any progressive CNS disorder (e.g., multiple sclerosis, CNS neoplasm) and evidence of acute intoxication or withdrawal, in the opinion of the study clinician.
* Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), HIV vaccine, systemic cytotoxic chemotherapy, or investigational therapy within 30 days prior to study entry.
* Currently breast-feeding.
* Requirement for any medications that have an absolute contraindication with any study drugs. In addition, we will exclude people taking rifampin.
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical illness.
* Prior use of nucleoside analogues, such as tenofovir, adefovir, or lamivudine, for treatment of hepatitis B for greater than 8 weeks while the subject was known to be HIV-infected.
* Any condition that, in the opinion of the investigators, would compromise the subject's ability to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-07; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Decline in neuropsychological performance at 96 weeks | 96 weeks
  Comparison of decline in NP performance between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Letendre, M.D., Principal Investigator — University of California, San Diego
Locations (2):
- China (2):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared in conference presentations and peer-reviewed publications. Data will also be made available on approval of requests for appropriate use.

REFERENCES:
- [Background] Heaton RK, Cysique LA, Jin H, Shi C, Yu X, Letendre S, Franklin DR, Ake C, Vigil O, Atkinson JH, Marcotte TD, Grant I, Wu Z; San Diego HIV Neurobehavioral Research Center Group. Neurobehavioral effects of human immunodeficiency virus infection among former plasma donors in rural China. J Neurovirol. 2008 Nov;14(6):536-49. doi: 10.1080/13550280802378880. PMID 18991068
- [Background] Cysique LA, Letendre SL, Ake C, Jin H, Franklin DR, Gupta S, Shi C, Yu X, Wu Z, Abramson IS, Grant I, Heaton RK; HIV Neurobehavioral Research Center group. Incidence and nature of cognitive decline over 1 year among HIV-infected former plasma donors in China. AIDS. 2010 Apr 24;24(7):983-90. doi: 10.1097/QAD.0b013e32833336c8. PMID 20299964
- [Background] Spector SA, Singh KK, Gupta S, Cystique LA, Jin H, Letendre S, Schrier R, Wu Z, Hong KX, Yu X, Shi C, Heaton RK; HNRC Group. APOE epsilon4 and MBL-2 O/O genotypes are associated with neurocognitive impairment in HIV-infected plasma donors. AIDS. 2010 Jun 19;24(10):1471-9. doi: 10.1097/QAD.0b013e328339e25c. PMID 20442634
- [Background] Letendre S, Marquie-Beck J, Capparelli E, Best B, Clifford D, Collier AC, Gelman BB, McArthur JC, McCutchan JA, Morgello S, Simpson D, Grant I, Ellis RJ; CHARTER Group. Validation of the CNS Penetration-Effectiveness rank for quantifying antiretroviral penetration into the central nervous system. Arch Neurol. 2008 Jan;65(1):65-70. doi: 10.1001/archneurol.2007.31. PMID 18195140
- [Background] Letendre SL, McCutchan JA, Childers ME, Woods SP, Lazzaretto D, Heaton RK, Grant I, Ellis RJ; HNRC Group. Enhancing antiretroviral therapy for human immunodeficiency virus cognitive disorders. Ann Neurol. 2004 Sep;56(3):416-23. doi: 10.1002/ana.20198. PMID 15349869
- See also: UCSD HIV Neurobehavioral Research Program — http://hnrc.hivresearch.ucsd.edu/
- See also: China Center for Disease Control and Prevention — http://www.chinacdc.cn
- See also: Beijing Youan Hospital — http://www.bjyah.com/en/index.asp
- See also: Beijing Ditan Hospital — http://www.bjditan.org/about_dicid_about_ditan_hospital.html